CLINICAL TRIAL: NCT02980770
Title: Postoperative Complications in Patients With Obesity Hypoventilation Syndrome Based on Base Excess- OHBE Study: A National, Multicenter, Observational Cohort Study
Brief Title: Postoperative Complications in Patients With Obesity Hypoventilation Syndrome
Acronym: OHBE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Collaborators: Elazig Education and Research Hospital (Unknown); Mustafa Kemal University (Other); Aydin Adnan Menderes University (Other); TC Erciyes University (Other); Sisli Hamidiye Etfal Training and Research Hospital (Other); Haydarpasa Numune Training and Research Hospital (Other); Fatih Sultan Mehmet Training and Research Hospital (Other); Konya Meram State Hospital (Other); Ankara City Hospital Bilkent (Other); Adana Numune Training and Research Hospital (Other Government); Tepecik Training and Research Hospital (Other); Sakarya University (Other); Ankara University (Other); Kahramanmaras Sutcu Imam University (Other); Trakya University (Other); Karadeniz Technical University (Other); Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government); Turkiye Yuksek Ihtisas Education and Research Hospital (Other Government); Ufuk University (Other); Kasımpasa Training and Research Hospital (Unknown); Nevsehir Public Hospital (Other Government); Hitit University (Other); Bulent Ecevit University (Other); Medipol University (Other)
Responsible Party: Sponsor
Other Study IDs: 70737436-050.06.04
Record Dates: First submitted 2016-11-30; First posted 2016-12-02 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Obstructive Sleep Apnea; Obesity Hypoventilation Syndrome; Hypercapnia; Post-Op Complication; Acid-Base Imbalance
Keywords: Obstructive Sleep Apnea; Obesity Hypoventilation Syndrome; Hypercapnia; Post-Op Complication; Acid-Base Imbalance
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity Hypoventilation Syndrome; Hypercapnia; Postoperative Complications; Acid-Base Imbalance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biochemistry, blood gases
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Obstructive Sleep Apnea (OSA): Patients with OSA
- Obesity-Hypoventilation Syndrome (OHS): Patients with OHS
- Normal Blood Gases: Normal Blood Gases

SUMMARY:
Obstructive sleep apnea (OSA) and Obesity-Hypoventilation Syndrome (OHS) are common conditions in obesity, which may influence the prognosis in patients undergoing surgery. There is a need for simple screening tools to identify such patients at high risk. The current multicenter observational study aims to investigate occurrence of OSA and OHS in obese individuals undergoing elective abdominal surgery and further address its impact on perioperative and postoperative complications.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) and Obesity-Hypoventilation Syndrome (OHS) are common conditions in obesity, which may influence the prognosis in patients undergoing surgery. There is a need for simple screening tools to identify such patients at high risk. The current multicenter observational study aims to investigate occurrence of OSA and OHS in obese individuals undergoing elective abdominal surgery by using questionnaires (STOPBANG questionnaire, Berlin Questionnaire, and Epworth Sleepiness Scale) and arterial blood gases. Perioperative and 72-h postoperative complications will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective abdominal surgery
* Body-Mass-Index >=30 kg/m2
* Ability to read and speak
* Signed informed consent.

Exclusion Criteria:

* Use of diuretics
* Use of theophylline
* Use of respiratory depressing drugs
* Severe lung disease (FEV1/FVC<%50)
* Severe hearth failure (EF<%35)
* Central nervous system or muscle disease
* Untreated hypothyroidism
* Renal failure (GFR<50)
* Total parenteral nutrition more than 72 hours
* Hypokalemia
* Hyponatremia
* Hypomagnesemia
* Hypoalbuminemia
* Known sleep apnea or obesity hypoventilation syndrome
* Blood transfusion from blood bank within 72 hours prior to surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive obese patients undergoing elective abdominal surgery
Sampling Method: Probability Sample
Enrollment: 999 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Cinel, Prof Dr, Study Chair — Marmara University Medical School
Locations (1):
- Marmara University Pendik Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No